CLINICAL TRIAL: NCT01002560
Title: Novel Prognostic Markers in Melanoma: a Protocol for the Analysis of Paraffin-embedded Tumour Samples
Brief Title: The Identification of Novel Prognostic Markers in Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Professor Martin Gore, Royal Marsden NHS Foundation Trust
Other Study IDs: CCR3078
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; Novel Prognostic Markers
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Malignant melanoma tumour tissue
- Benign pigmented lesions & other skin cancers: Normal skin, benign melanocytic tumours, and skin cancers from lineages other than melanocytic, to be used as negative controls

SUMMARY:
The purpose of this project is to analyze tumour tissue from a group of subjects with malignant melanoma, who have been treated at the Royal Marsden Hospital.

DETAILED DESCRIPTION:
Background - The Royal Marsden Hospital and the Institute of Cancer Research constitute the largest comprehensive cancer centre in Europe. In addition to an in-house drug development program, phase I - phase III clinical trials of novel anti-cancer agents are hosted. In order to investigate the optimal use of novel molecularly targeted agents, access to clinical tumour samples is needed in order to determine which particular cancer type expresses a molecular "signature" that may indicate potential therapeutic utility. Understanding such signatures should accelerate the registration of new drugs for routine cancer therapy; offering the potential of selecting those patients with tumour types most likely to benefit from therapy. Furthermore, new insights into disease biology may be gained.

Main research question/ objective - Are there features of primary melanoma or lymph node metastases that predict subsequent clinical outcome better than existing markers?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of melanoma
* Adequate paraffin-embedded material available for analysis.
* Adequate clinical follow-up information
* Written informed consent where applicable

Exclusion Criteria:

* Inadequate paraffin-embedded material available
* Inadequate clinical follow-up information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group of subjects with malignant melanoma, who have been treated at the Royal Marsden Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Given that the nature of the research is qualitative, there is no primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Martin Gore, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom